CLINICAL TRIAL: NCT02309268
Title: LARIAT: Atrial Appendage Closure Prospective Observational Study
Brief Title: Atrial Appendage Closure Prospective Observational Study
Acronym: LARIAT
Status: Withdrawn | Type: Observational
Why Stopped: The principal linvestigator decided not to continue the registry. No patient were enrolled. CLosure to the registry was done October 2014
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: LARIAT
Record Dates: First submitted 2014-08-01; First posted 2014-12-05 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Closure
Keywords: left atrial appendage closure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research is to monitor how well patients do after surgery for treatment of left atrial appendage (LAA).

DETAILED DESCRIPTION:
Patients will be followed in an observational study. We propose to do a single follow-up TEE at 3 to 6 months (this is standard of care) to confirm LAA (left atrial appendage) occlusion. The TEE is not mandatory (this is not a clinical trial), but will be strongly recommended to patients to confirm the efficacy of treatment. This will help confirm whether patients may safely remain off anticoagulation. The risks of TEE are a less than 1 in 1000 risk of death, and a 1% or less risk of a major complication, such as esophageal perforation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Atrial fibrillation
* Are poor candidates to take warfarin
* Have elected to undergo a LARIAT procedure

Exclusion Criteria:

* none

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being asked to take part in this study have a heart disorder known as atrial fibrillation (AF) and are poor candidates to take blood thinning drug known as warfarin (Coumadin), and have elected to undergo LARIAT procedure.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Clinical Progress | At regular visits ( 3 months and annually)
  Patients who agree to participate in the registry will allow the Investigators to document their clinical progress and compare their progress to other participants in the study. Meanwhile, the patient will continue to receive routine care from their physician, just as they would if they did not participate in the study. Any information published as a result of this registry, will be kept anonymous. There is no known risk in participating in this study as it is only an observational study.

CONTACTS AND LOCATIONS:
Overall Officials: kenneth A Ellenbogen, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Medical Center, Richmond, Virginia, United States